CLINICAL TRIAL: NCT07332546
Title: External Oblique Intercostal Block for Postoperative Pain After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: EOIB for Pain After Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shiyou Wei (Other)
Responsible Party: Sponsor-Investigator, Shiyou Wei, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250322
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Laparoscopic Cholecystectomy
Keywords: External oblique intercostal block; Ultrasonography, Interventional; Nerve Block; Quality of recovery (QoR-15)
MeSH Terms: conditions — Pain, Postoperative | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to one of two parallel groups: bilateral ultrasound-guided external oblique intercostal block (EOIB) or control (no regional block). Each participant receives only the assigned intervention.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to group assignment. Participants and clinical care providers/investigators are not blinded because the control group does not receive a regional block.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOIB Group (Experimental): Participants receive bilateral ultrasound-guided external oblique intercostal block (EOIB) (15 mL of the study local anesthetic mixture per side) in addition to standard general anesthesia and standardized postoperative analgesia (IV PCA butorphanol ).
  Interventions: Other: External oblique intercostal block (EOIB)
- Control Group (Sham Comparator): Participants do not receive any regional block. They receive standard general anesthesia and standardized postoperative analgesia only (IV PCA butorphanol).
  Interventions: Other: Standard care without regional block

INTERVENTIONS:
Other: External oblique intercostal block (EOIB) — Bilateral ultrasound-guided external oblique intercostal block performed under sterile conditions after induction of general anesthesia and before surgical incision. Using an in-plane technique, the block is performed at the level of the 6th rib in the 6th-7th intercostal space. A local anesthetic mixture is injected with a total volume of 15 mL per side (prepared by mixing 0.75% ropivacaine with normal saline).
  Arms: EOIB Group
Other: Standard care without regional block — Participants do not receive any regional anesthesia/nerve block (including external oblique intercostal block). All participants receive standard general anesthesia and the same standardized postoperative multimodal analgesia regimen as per protocol, including intravenous patient-controlled analgesia (PCA) with butorphanol.
  Arms: Control Group

SUMMARY:
This prospective, randomized, controlled, assessor-blinded trial will evaluate whether bilateral ultrasound-guided external oblique intercostal block (EOIB) reduces postoperative opioid consumption and improves pain control after laparoscopic cholecystectomy, compared with no block.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is a common procedure, yet postoperative pain remains clinically significant despite routine multimodal analgesia, and opioid use may cause adverse effects. External oblique intercostal block (EOIB) is a newer ultrasound-guided fascial plane block that may provide effective analgesia for upper abdominal surgery.

This study is a prospective, randomized, controlled, assessor-blinded trial in patients undergoing elective laparoscopic cholecystectomy. A total of 56 participants will be randomized 1:1 to receive either bilateral ultrasound-guided EOIB or no regional block. EOIB will be performed bilaterally under ultrasound guidance at the level of the 6th rib in the 6th-7th intercostal space using an in-plane technique, with 15 mL of study local anesthetic mixture injected per side. Postoperatively, all participants will receive standardized multimodal analgesia, including intravenous patient-controlled analgesia (PCA) with butorphanol and non-opioid analgesics per protocol.

The primary outcome is total opioid consumption during the first 24 hours after surgery. Secondary outcomes include postoperative pain scores (VRS) at prespecified time points, quality of recovery (QoR-15) at 24 hours, opioid consumption from 24-48 hours, postoperative nausea and vomiting, intraoperative hemodynamic events, time to first flatus, and length of hospital stay. The trial aims to determine whether adding bilateral EOIB to standard analgesia can reduce opioid requirements and improve recovery after laparoscopic cholecystectomy.

Note for your protocol alignment: your document contains a potential inconsistency about "no other opioids within 72 hours" versus recording "rescue opioid" use; you may want to standardize this wording before final submission.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85 years, regardless of gender
* American Society of Anesthesiologists (ASA) physical status classification I-III
* Scheduled for elective laparoscopic cholecystectomy
* Ability to use the intravenous patient-controlled analgesia (IV PCA) system

Exclusion Criteria:

* Hepatic disease (e.g., liver enzyme levels ≥ 2× the upper limit of normal)
* Renal disease (e.g., serum creatinine levels ≥ 2× the upper limit of normal)
* Allergy or known hypersensitivity to local anesthetics
* Females who are pregnant or lactating
* Conversion to open surgery
* Coagulopathy or current use of anticoagulant medications
* Opioid use for more than 2 weeks in the past 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Total Butorphanolconsumption in the first 24 hours after surgery | 0-24 hours after surgery
  Total Butorphanol consumption during the first 24 hours postoperatively. A relative difference of 30% is considered clinically significant.

SECONDARY OUTCOMES:
Pain score (VRS) at 24 hours after surgery | 24 hours after surgery
  Postoperative pain intensity measured using the Verbal Rating Scale (VRS; 0 = no pain, 10 = worst pain imaginable) at 24 hours after surgery.
Quality of recovery at 24 hours (QoR-15 score) | 24 hours after surgery
  Quality of recovery assessed using the 15-item Quality of Recovery questionnaire (QoR-15); total score at 24 hours postoperatively.
Butorphanol consumption from 24 to 48 hours after surgery | 24-48 hours after surgery
  Total butorphanol consumption recorded during postoperative hours 24-48 (including PCA-delivered dose and any additional butorphanol administered).
Pain score (VRS) at 48 and 72 hours after surgery | 48 hours and 72 hours after surgery
  Postoperative pain intensity measured using the Verbal Rating Scale (VRS; 0-10) at 48 hours and 72 hours after surgery.
Incidence of postoperative nausea and vomiting within 72 hours | 1-6 hours, 7-24 hours, 25-48 hours, and 49-72 hours after surgery (up to 72 hours)
  Incidence of nausea and/or vomiting recorded during postoperative time intervals (1-6 h, 7-24 h, 25-48 h, and 49-72 h); summarized up to 72 hours.
Incidence of intraoperative hypotension and hypertension | Intraoperative period
  Incidence of intraoperative hypotension and intraoperative hypertension during surgery, recorded per protocol definitions. Blood pressure increase exceeding 30% of the baseline value is used as the measurement criterion.
Time to first flatus | Within 3 days after surgery
  Time from the end of surgery to the first passage of flatus.
Postoperative length of hospital stay | Within 7 days after surgery
  Duration of hospital stay after surgery, measured from the time of surgery to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lv, PhD, Study Chair — Shanghai Pulmonary Hospital, Tongji University, Shanghai, China
Locations (1):
- Tianmen First People's Hospital, Tianmen, Hubei, China

IPD SHARING:
Plan to Share IPD: No